CLINICAL TRIAL: NCT06932952
Title: A Dose Escalation and Expansion Trial With the SIRPα-directed Monoclonal Antibody BYON4228 Alone and in Combination to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics and Efficacy in Patients With Advanced or Metastatic Solid Tumors
Brief Title: A Dose Escalation and Expansion Trial With BYON4228 Alone and in Combination in Patients With Advanced or Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Byondis B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BYON4228.002; 2024-517952-37-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor
Keywords: mAB; Monoclonal antibody; SIRPα; CD47; SIRP
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BYON4228 + Pembrolizumab (Experimental)
  Interventions: Drug: BYON4228 + Pembrolizumab

INTERVENTIONS:
Drug: BYON4228 + Pembrolizumab — BYON4228 is a humanized monoclonal antibody (mAb) directed against SIRPα. BYON4228 IV infusion every three weeks until disease progression or unacceptable toxicity. Different doses. Pembrolizumab IV infusion (200 mg) every three weeks from the second treatment cycle onwards.

SUMMARY:
This is a phase I trial with BYON4228, a humanized monoclonal antibody (mAb) directed against signal regulatory protein (SIRP)α in solid tumors, alone and in combination with pembrolizumab.

DETAILED DESCRIPTION:
This study includes a dose escalation part (Part 1) in which the MTD or OBD and RDE(s) will be determined. This trial includes an expansion part (Part 2) to evaluate efficacy and safety of BYON4228 in combination with pembrolizumab in specific patient cohorts.

BYON4228 is a humanized IgG1 mAb directed against SIRPα. BYON4228 binds SIRPα expressed on innate immune cells, especially monocytes, macrophages and neutrophils. BYON4228 blocks binding of SIRPα to CD47 and inhibits signaling through the CD47-SIRPα axis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically confirmed, locally advanced or metastatic cancer who has progressed on standard therapy or for whom no standard therapy exists:

  * Part 1 (dose escalation): Solid tumors of any origin;
  * Part 2 (expansion): Patients with other solid tumor types indicated for pembrolizumab monotherapy;
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1;
* For Part 2 only: at least one measurable cancer lesion as defined by the Response Evaluation Criteria for Solid Tumors (RECIST version 1.1);
* Adequate baseline organ function.

Exclusion Criteria:

* Having been treated with CD47 or SIRPα targeting agents or other anticancer therapy within 4 weeks prior to the start of IMP treatment;
* History of hypersensitivity or allergic reaction to any of the excipients of BYON4228;
* Any contraindication to pembrolizumab treatment;
* For Part 2: Patients previously given a PD-1 or PD-L1 inhibitor who had subsequent disease progression within 8 weeks of initiation;
* Symptomatic brain metastases;
* History of autoimmune disorders;
* Severe active infection or other severe uncontrolled systemic disease;
* Having clinically significant cardiovascular disease;
* Known infection of Hepatitis B, C or E.

Key inclusion and exclusion criteria details are listed here, additional requirements may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities | 21 days
Objective Response Rate | 2 years
  Part 2 (expansion): To evaluate the objective tumor response rate (ORR).

CONTACTS AND LOCATIONS:
Locations (6):
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - UZ Leuven, Leuven
- Spain (2):
  - CIOCC Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester
  - The Royal Marsden, Sutton